CLINICAL TRIAL: NCT07390513
Title: Electrophysiological Outcomes After Transcatheter Aortic Valve Replacement
Acronym: TAVR-ELECTRO
Status: Active, not recruiting | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Pan Xiangbin, Professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2024-2428; NCRC2020009 (Other Grant/Funding Number: National Clinical Research Center for Cardiovascular Diseases, Fuwai Hospital, Chinese Academy of Medical Sciences)
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Aortic Valve Stenosis; Arrhythmia
MeSH Terms: conditions — Aortic Valve Stenosis; Arrhythmias, Cardiac | interventions — Clopidogrel

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: TAVR Aspirin and clopidogrel — This is an observational registry study. All participants undergo transcatheter aortic valve replacement (TAVR) as part of standard clinical care for severe aortic stenosis. The choice of valve type (balloon-expandable or self-expanding), valve brand, valve size, access route, and peri-procedural management strategies are determined by the local heart team according to current clinical guidelines and routine practice.
  No additional investigational intervention is mandated by the registry protocol. The study does not alter clinical decision-making, procedural techniques, or post-procedural treatment strategies. Instead, the registry systematically collects clinical, echocardiographic, electrocardiographic, and procedural data before and after TAVR to evaluate electrophysiological outcomes.
  Post-procedural rhythm assessment, including standard electrocardiography and ambulatory electrocardiographic monitoring, is performed as part of routine follow-up care. Data on ventricular arrhythm

SUMMARY:
The TAVR-ELECTRO Registry (Electrophysiological Outcomes After Transcatheter Aortic Valve Replacement) is a single-center, observational cohort study designed to systematically evaluate the occurrence, temporal evolution, and determinants of cardiac arrhythmias following transcatheter aortic valve replacement (TAVR) in patients with severe aortic stenosis.

This registry retrospectively enrolls consecutive patients undergoing TAVR at Fuwai Hospital, Chinese Academy of Medical Sciences, and collects comprehensive clinical, echocardiographic, electrocardiographic, and procedural data. Particular emphasis is placed on post-procedural electrophysiological outcomes, including ventricular arrhythmias, atrial arrhythmias, and conduction disturbances. Serial rhythm assessments using standard electrocardiography and ambulatory electrocardiographic monitoring are performed during follow-up to characterize arrhythmic burden and its dynamic changes over time.

The primary objective of the TAVR-ELECTRO Registry is to identify clinical, haemodynamic, and procedural factors associated with post-TAVR arrhythmic outcomes and recovery patterns, thereby improving the understanding of electrophysiological remodeling after TAVR and informing post-procedural risk stratification and management strategies.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years at the time of transcatheter aortic valve replacement (TAVR). Diagnosis of severe aortic stenosis based on current guideline-recommended echocardiographic criteria.

Undergoing transcatheter aortic valve replacement (TAVR) as part of routine clinical care.

Availability of baseline electrocardiographic assessment, including ambulatory electrocardiographic monitoring for evaluation of premature ventricular contraction (PVC) burden.

Completion of post-procedural rhythm follow-up, including ambulatory electrocardiographic monitoring at 12 months after TAVR.

Ability to provide informed consent or availability of legally authorized consent, as required by the institutional review board.

Exclusion Criteria:

Absence of premature ventricular contractions at baseline (PVC burden = 0), as PVC response cannot be meaningfully assessed in this population.

Presence of a permanent pacemaker or implantable cardioverter-defibrillator prior to TAVR.

Receipt of catheter ablation for atrial or ventricular arrhythmias before TAVR or during the follow-up period.

Death occurring during the index hospitalization or before completion of rhythm follow-up.

Inability to complete scheduled electrocardiographic or ambulatory rhythm assessments during follow-up.

Missing or incomplete key electrocardiographic, echocardiographic, or follow-up data required for outcome assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients with severe aortic stenosis who undergo transcatheter aortic valve replacement (TAVR) as part of routine clinical care at Fuwai Hospital, Chinese Academy of Medical Sciences. Eligible participants include consecutive patients who receive TAVR and undergo systematic post-procedural rhythm evaluation as part of standard follow-up.
  The registry focuses on patients with available baseline and follow-up electrocardiographic assessments, allowing for longitudinal evaluation of cardiac arrhythmias after TAVR. Particular attention is given to ventricular arrhythmias, including premature ventricular contractions, as well as atrial arrhythmias and conduction disturbances occurring during follow-up.
  This study population reflects a real-world cohort of patients treated with contemporary TAVR devices and management strategies, providing comprehensive clinical, echocardiographic, electrocardiographic, and procedural data to characterize electrophysi
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Premature Ventricular Contraction (PVC) Response at 12-Month Follow-up | Baseline to 12 months after transcatheter aortic valve replacement (TAVR)
  PVC response is defined as a reduction of ≥50% in premature ventricular contraction burden at 12 months compared with baseline. PVC burden is quantified as the total number of premature ventricular contractions per 24 hours, assessed by 24-hour ambulatory electrocardiographic monitoring. Patients without detectable PVCs at baseline are excluded from the primary responder analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- National Clinical Research Center for Cardiovascular Diseases, Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No